CLINICAL TRIAL: NCT04927676
Title: Hormone Profile in Women With Hypogonadotropic Hypogonadism - a Prospective Pilot Study
Brief Title: Hormones in Hypogonadotropic Hypogonadism
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Principal Investigator, Johannes Ott, Associate Professor, Consultant Physician, Medical University of Vienna
Other Study IDs: 2802/2021
Record Dates: First submitted 2021-05-31; First posted 2021-06-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: AMH; Hypogonadism, Hypogonadotropic; Follicle Cyst
MeSH Terms: conditions — Hypogonadism; Follicular Cyst | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples taken as part of routine clinical practice, including hormone status: AMH, FSH, LH, Estradiol, SHBG, DHEAS, Testosterone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — Blood samples were taken from a peripheral vein as part of clinical routine. Subsequently, a hormone status is determined.

SUMMARY:
Therefore, the main objective of this prospective pilot study is to evaluate a complete hormonal profile in women with hypogonadotropic hypogonadism, including anti-mullerian hormone (AMH) and antral follicle count. Changes in this regard will be evaluated after 2 months of individual treatment.

DETAILED DESCRIPTION:
The objective of this prospective cohort pilot study is to evaluate a complete hormonal profile including AMH and antral follicle count in women with hypogonadotropic hypogonadism (HH). As a secondary study objective, changes in these two parameters will be examined after 2 months of individual treatment. The data collected will be used to plan future studies in the field.

The primary hypothesis is, that AMH levels which range from 0.5 ng/mL to 7.0 ng/mL and antral follicular counts which range from 2 to 20 can be found in women with HH.

As secondary hypothesis the investigators assume that the AMH levels and the antral follicular counts of women with HH do not change within two months of treatment with estrogen-/gestagen-replacement therapy or no treatment, whereas AMH levels and antral follicular counts will increase significantly after two months of pulsatile gonadotropin-releasing hormone (GnRH) treatment.

Primary outcome parameters are serum level of AMH and the antral follicular count. Secondary outcome parameters as for the descriptive analysis are: follicle stimulating hormone (FSH), luteinizing hormone (LH), estradiol (either during amenorrhea or on cycle day 2-5 in the course of treatment), sexual hormone binding globulin (SHBG), testosterone, dehydroepiandrosterone-sulfate (DHEAS), results of a Dual Energy X-ray Absorptiometry (DEXA; if performed), duration since last normal menstruation, patient's age and body mass index (BMI).

The following parameters will be collected and included in the database. They do not require additional effort on behalf of the patients. All data will be obtained using the study-specific case report form and will be entered into a SPSS (IBM SPSS Statistics Software) database in a semi-anonymized manner: Patient's age, Body mass index, duration since last normal menstruation, FSH, LH, Estradiol, SHBG, Testosterone, DHEAS, DEXA results, AMH, Antral follicular count. Data acquisition will be conducted to give an exact characterization of the patient population to allow a comparison with the published literature. All taken blood samples are performed as part of the clinical routine at the Clinical Institute of Laboratory Medicine at Vienna General Hospital.

The study is designed as a pilot study. This is due to the lack of sufficient literature on this topic. Fifty women with HH and secondary amenorrhea will be included.

Potential participants are informed about the procedure, clinical relevance and the balance of risk and benefits incurred through study participation. Patients willing to participate will express this through written affirmation (a "consent form").

All above mentioned data are numerical data and will be reported as mean and standard deviations. Differences between different treatment groups will be tested using unpaired t-tests, whereas differences within groups (baseline to follow-up examinations) will be tested using paired t-tests. Statistical analyses were performed with SPSS 26.0. P-values <0.05 will be considered statistically significant.

Extreme values will be double-checked. In addition, random checks by two independent investigators will be conducted to ensure the accuracy of the data.

In this prospective study, no further data acquisitions, follow-up examinations or surveys will be necessary. Accordingly, if patients would be undergoing the described interventions (blood retrieval, DEXA analysis) independent of their choice to participate, this should not shift cost or risk for them. The analysis and publication of the data will be done with patient de-identification.

The decision on how to proceed after the initial diagnosis is made in the course of routine clinical practice, after the medical team in charge of the patient has provided precise information on the advantages and risks of the respective procedures. Participation in the study therefore has no influence on the type of further procedure or therapy.

The study is conducted as independent official research. The company "Ferring Arzneimittel GmbH (Gesellschaft mit beschränkter Haftung)" is supporting the conduct of the study with 3,000 euros. The company produces the preparation "LutreLef", which is administered to some patients as part of the clinical routine with the pump system "LutrePulse".

ELIGIBILITY:
Inclusion Criteria:

* Patient with HH and secondary amenorrhea. HH is defined as absence of spontaneous menstruation for ≥6 months, no abrupt menstrual bleeding after progesterone therapy, and normal or low serum FSH and LH levels.
* The patient gave written informed consent to the study after receiving detailed information and education from medical contributors at the Department of Obstetrics and Gynecology, Medical University of Vienna.
* Age between >18 and <35 years.

Exclusion Criteria:

* Latent or manifest hypothyroidism (TSH >4 micromole/milliliter) or current thyroid hormone replacement therapy.
* No existing informed consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with HH and secondary amenorrhea presenting to the Department of Obstetrics and Gynecology, Medical University of Vienna. The target number of cases for this pilot study is 50 patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
AMH | 2 months
  Evaluation of a complete hormone profile including AMH in women with HH
antral follicle count | 2 months
  Evaluation of the antral follicle count in women with HH

SECONDARY OUTCOMES:
AMH after 2 months | 2 months
  Changes in this parameter studied after 2 months of individual treatment (after starting estrogen/progestin replacement therapy or without treatment)
Antral follicle count after 2 months | 2 months
  Changes in this parameter studied after 2 months of individual treatment (after starting estrogen/progestin replacement therapy or without treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ott, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No